CLINICAL TRIAL: NCT07130968
Title: Real-World Cohort Study of Cardiopulmonary Function in Chinese Patients With Cardiovascular Disease: CPET Evaluation and Five-Year Prognostic Follow-Up Based on a Multicenter Structured Data Platform
Acronym: China-CPET
Status: Enrolling by invitation | Type: Observational
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: Yuebei People's Hospital (Other); People's Hospital of Xinjiang Uygur Autonomous Region (Other); Gansu Provincial Hospital (Other); Shenzhen Center for Chronic Disease Control (Other); Yangjiang People's Hospital (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); Nanfang Hospital, Southern Medical University (Other); Qingdao Municipal Hospital (Other); Weifang People's Hospital (Other); Guangming District People's Hospital of Shenzhen (Unknown)
Responsible Party: Principal Investigator, Huan Ma, Deputy Director of Cardiology, Director of the Department of Cardiac Rehabilitation, Guangdong Provincial People's Hospital
Other Study IDs: KY2025-499-03
Record Dates: First submitted 2025-08-13; First posted 2025-08-19 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: MACE; Cardiac Death; Unplanned Repeat Revascularization; Cardiac Rehospitalization; Non-fatal Myocardial Infarction; Stroke
Keywords: Cardiopulmonary Exercise Testing; Cardiovascular Diseases; Major Adverse Cardiovascular Events (MACE); Prognosis; Exercise Capacity; Cardiorespiratory Fitness; Clinical Outcomes; Real-world Study
MeSH Terms: conditions — Death; Stroke; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cardiovascular disease patient with MACE: cardiovascular disease patient with MACE（Cardiac death, unplanned revascularization, cardiac readmission, non-fatal myocardial infarction, and stroke）
- cardiovascular disease patient without MACE

SUMMARY:
The goal of this observational study is to observe the characteristics of cardiopulmonary exercise testing (CPET) parameters in patients across different cardiovascular diseases and to evaluate the predictive value of multiparameter cardiopulmonary indices for 5-year major adverse cardiovascular events (MACE).

DETAILED DESCRIPTION:
To investigate the CPET characteristics in patients with various cardiovascular diseases (including acute myocardial infarction, heart failure, cardiomyopathy, valvular heart disease, coronary artery disease, and perioperative cardiac surgery), with annual follow-up of major adverse cardiovascular events (MACE) for five years, and to establish the predictive value of combined CPET parameters for MACE in this population

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-80 years,
2. Ability to comprehend and provide written informed consent.

Exclusion Criteria:

1. Comorbid severe conditions (e.g., recent acute myocardial infarction, unstable angina, uncontrolled arrhythmias, severe aortic coarctation or descending aortic aneurysm, acute myocarditis or pericarditis, acute congestive heart failure, acute respiratory failure, resting oxygen saturation <93%, recent arterial or pulmonary embolism, pulmonary edema).
2. Conditions potentially exacerbated by exercise (e.g., acute cardiac insufficiency, exercise-induced asthma, epilepsy).
3. Physical disability due to musculoskeletal or neuromuscular disorders.
4. Pregnancy or lactation.
5. Patients deemed unsuitable for participation by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: China CardioVascular Disease Patient and healthy control group
Sampling Method: Non-Probability Sample
Enrollment: 200000 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2035-12-30 (Estimated); Study Completion 2035-12-30 (Estimated)

PRIMARY OUTCOMES:
Characteristics of CPET parameters across different cardiovascular diseases. | After enrollment
  Cardiopulmonary exercise testing (CPET) was performed using exercise cardiopulmonary testing systems from VYAIRE (Germany) and SCHILLER (Switzerland). A symptom-limited maximal exercise test with a 1-minute ramp incremental protocol (Ramp protocol) was adopted, designed to complete the workload test within 8-12 minutes according to the incremental power calculation formula.
  The incremental workload was calculated as follows:
  Unloaded VO₂ (ml/min) per minute = 150 + (6 × body weight) Predicted peak VO₂max (ml/min) per minute for males = (height in cm - age in years) × 20 Predicted peak VO₂max (ml/min) per minute for females = (height in cm - age in years) × 14 Incremental power per minute = (predicted peak VO₂max - unloaded VO₂)/100
  During exercise, real-time cardiopulmonary parameters were collected, including peak oxygen uptake (VO₂peak), anaerobic threshold (AT), maximal cycling workload, respiratory rate, minute ventilation (VE), and ventilatory efficiency, among others.
Incidence of 5-year MACE | from enrollment to 5 years post-enrollment
  MACE (cardiovascular death, unplanned repeat revascularization, cardiac rehospitalization, non-fatal myocardial infarction, stroke)

SECONDARY OUTCOMES:
Incidence of individual events of MACE per year (incidence of cardiac death, unplanned rereconstitution, cardiac rehospitalization, nonfatal myocardial infarction, and stroke) | yearly for 5 years (Year 1/2/3/4/5 from enrollment)

OTHER OUTCOMES:
Incidence rate of adverse events during exercise | During each exercise session and within 24 hours after exercise

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shephard RJ, Balady GJ. Exercise as cardiovascular therapy. Circulation. 1999 Feb 23;99(7):963-72. doi: 10.1161/01.cir.99.7.963. No abstract available. PMID 10027821
- [Result] Fiuza-Luces C, Santos-Lozano A, Joyner M, Carrera-Bastos P, Picazo O, Zugaza JL, Izquierdo M, Ruilope LM, Lucia A. Exercise benefits in cardiovascular disease: beyond attenuation of traditional risk factors. Nat Rev Cardiol. 2018 Dec;15(12):731-743. doi: 10.1038/s41569-018-0065-1. PMID 30115967
- [Result] DeCato TW, Haverkamp H, Hegewald MJ. Cardiopulmonary Exercise Testing (CPET). Am J Respir Crit Care Med. 2020 Jan 1;201(1):P1-P2. doi: 10.1164/rccm.2011P1. No abstract available. PMID 31891317
- See also: websites associated with the cited references — https://pubmed.ncbi.nlm.nih.gov/30115967/